CLINICAL TRIAL: NCT05409742
Title: Masseter Muscle Activity and Post-Operative Pain in A Group of Egyptian Children With Carious Primary Molars Treated With Hall Vs Modified Hall Technique: A Randomised Clinical Trial
Brief Title: Masseter Muscle Activity and Post-operative Pain in a Group of Egyptian Children Treated With Hall Technique Vs Modified Hall Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Abdelazim Abdelsayed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PEDO 4-8-3
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Masseter Muscle Activity
Keywords: Hall technique; Modified Hall technique; Stainless steel crowns

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Hall technique (Active Comparator)
  Interventions: Diagnostic Test: Modified Hall technique
- Hall Technique (Experimental)
  Interventions: Diagnostic Test: Modified Hall technique

INTERVENTIONS:
Diagnostic Test: Modified Hall technique — The standard Hall technique was later modified with several modifications including occasional/rare use of anesthetic and about 1 mm proximal slice that the preformed metal crown fits without separation, and minimal occlusal reduction of the cusps

SUMMARY:
The study aims to evaluate postoperative pain and masseter muscle activity in a group of Egyptian children with carious primary molars treated with Hall Vs modified Hall Technique (with proximal and occlusal reduction).

ELIGIBILITY:
Inclusion Criteria:

* Children 5-7 years with carious lower second primary molars
* Both genders.
* Systemically and mentally healthy.

Exclusion Criteria:

* History of systemic or mental conditions.
* Special health care needs who require pharmacological management before dental treatment.
* Acute dental pain or trauma.
* Extremely uncooperative children who require being treated under general anesthesia.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Masseter muscle activity measured by Electromyograph | 6 weeks
  muscle activity will be measured following the cementation of the crown

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo University, Cairo, EL-Manial, Egypt